CLINICAL TRIAL: NCT00217945
Title: Does Shared Decision-Making Improve Adherence in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 294; R01HL069358 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Lung Diseases; Asthma
MeSH Terms: conditions — Lung Diseases; Asthma

INTERVENTIONS:
Behavioral: Shared-Decision Making

SUMMARY:
To evaluate a model of shared decision-making for asthma treatment, appropriate to the needs of African American, Latino, Chinese, and other Asian and low income Caucasian patients to adherence to asthma controller medications in a two-year randomized clinical trial in 302 minority and low-income adults, 18-70 years of age, with suboptimally controlled, persistent asthma, paralleling a simultaneous evaluation being conducted in 311 Caucasian and Asian/Pacific Island adults, (total n=613), and to examine psychological mechanisms mediating the effects of the intervention on adherence and of adherence on asthma outcomes.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is a chronic inflammatory disorder of the airways. Despite major advances in understanding of its pathophysiology and management, asthma outcomes have not shown parallel improvement. Many patients with asthma are poorly controlled and have sub-optimal health status. Asthma care management by a trained non-physician health professional has developed as a means of addressing the problems of patients evidencing poor control and/or poor adherence to controller medications. Shared decision making (SDM) between clinician and patient has also been proposed as a means of getting greater patient involvement in their care, with the idea that this may improve medication adherence and outcomes. However, significant patient involvement also might result in less adequate regimens than would management based on guidelines (MBG). Even so, increased adherence to a less adequate regimen might result in better outcomes than poor adherence to an optimal regimen.

DESIGN NARRATIVE:

Better Outcomes of Asthma Treatment (BOAT) is a randomized controlled trial (a collaborative study designed to compare the effectiveness of three strategies for managing patients, 18-70 years of age, with suboptimally controlled, persistent asthma. The three treatment strategies are: usual care (UC); management by guidelines (MG); and a third, shared decision making (SDM) arm, that seeks to formally involve the patient in the therapeutic decision-making process. Under the present grant, 302 study participants were recruited from the membership of the Kaiser Permanente - Northern California Region (KPNC), San Francisco, Oakland, and Richmond medical centers. In the collaborating grant (No.HL67092-03) 311 patients were recruited from Kaiser Permanente clinical facilities in Portland, OR, and Honolulu, HI. Patients were randomized equally to the three treatment arms following baseline assessment of asthma control, medication use, lung function, and other behavioral and psychological characteristics. Their health care utilization for asthma and acquisition of asthma medications is being followed for a total of 24 months post-randomization through health system records, and they are being reassessed at 12 mos. Those assigned to the care management conditions received asthma education and objective feedback on their level of asthma control. Those assigned to the MBG condition were prescribed a regimen appropriate to the severity of their asthma in accordance with standard guidelines for asthma management. Those assigned to the SDM condition participated in a process to elicit their goals for their asthma treatment and their priorities regarding their asthma medications, and then engaged in a process of shared decision making with the care manager designed to arrive at a prescribed regimen that satisfied their goals and preferences. Analysis of the data will compare the two care management approaches with usual care and with each other in terms of the primary outcomes.

ELIGIBILITY:
* Kaiser Health Care Program member for more than 1 yr.
* Site: Portland, OR, Honolulu, HI, San Francisco, Oakland, or Richmond, CA.
* Confirmed diagnosis of persistent asthma with currently prescribed medications; no daily or alternate daily oral corticosteroid
* Evidence of poorly controlled asthma: score of >=1 on ATAQ asthma control questionnaire1 and either overuse of rescue medication vs. controller medications and/or recent emergency visit or hospitalization for asthma
* COPD not the primary lung disease diagnosis
* Regular use of Inhaled Corticosteroid (ICS) and current/ex-smokers: >= 8% increase in FEV1 post-bronchodilator; if no routine ICS use +/- smoking HX: >= 12% increase required; non-smokers using ICS regularly not required to reverse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Wilson — Palo Alto Medical Foundation

REFERENCES:
- [Background] Wilson SR, Buist AS, Holup J, Brown NL, Lapidus J, Luna V, Verghese S. Shared Decision Making vs. Management by Guidelines: Impact on Medication Regimen. Poster presented at the 2005 Annual Meeting of the American Thoracic Society, San Diago, CA, May 24, 2005. Proceedings of the American Thoracic Society; Vol.2 Abstracts Issue; 2005.
- [Derived] Wilson SR, Strub P, Buist AS, Knowles SB, Lavori PW, Lapidus J, Vollmer WM; Better Outcomes of Asthma Treatment (BOAT) Study Group. Shared treatment decision making improves adherence and outcomes in poorly controlled asthma. Am J Respir Crit Care Med. 2010 Mar 15;181(6):566-77. doi: 10.1164/rccm.200906-0907OC. Epub 2009 Dec 17. PMID 20019345